CLINICAL TRIAL: NCT07324200
Title: Objective Assessment of Intraocular Lens Tilt and Decentration
Status: Not yet recruiting | Type: Observational
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MDEV113OCTI
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Tilt and Decentration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- TECNIS refractive non-toric IOL models: The primary objective of this study is to evaluate the repeatability and reproducibility (R&R) of a method based on Optical Coherence Tomography (OCT) image analysis for assessing IOL tilt and decentration in patients unilaterally or bilaterally implanted with TECNIS refractive non-toric IOL models.
  Interventions: Diagnostic Test: OCT Imaging Test
- TECNIS diffractive non-toric IOL models: The primary objective of this study is to evaluate the repeatability and reproducibility (R&R) of a method based on Optical Coherence Tomography (OCT) image analysis for assessing IOL tilt and decentration in patients unilaterally or bilaterally implanted with TECNIS diffractive non-toric IOL models.

INTERVENTIONS:
Diagnostic Test: OCT Imaging Test — The primary objective of this study is to evaluate the repeatability and reproducibility (R&R) of a method based on Optical Coherence Tomography (OCT) image analysis for assessing IOL tilt and decentration in patients unilaterally or bilaterally implanted with TECNIS refractive or diffractive non-toric IOL models.
  Other Names: Basic Science
  Groups: TECNIS refractive non-toric IOL models

SUMMARY:
Prospective, multi-center, non-interventional, open label, randomized clinical study.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the repeatability and reproducibility (R&R) of a method based on Optical Coherence Tomography (OCT) image analysis for assessing IOL tilt and decentration in patients unilaterally or bilaterally implanted with TECNIS refractive or diffractive non-toric IOL models.

ELIGIBILITY:
INCLUSION CRITERIA (ALL CRITERIA APPLY TO STUDY EYE)

1. Read, understand, and sign the informed consent and HIPAA authorization forms, and receive a fully executed copy of the signed forms.
2. Appear capable and willing to adhere to the clinical protocol instructions.
3. Be 22 years of age or older at the time of screening.
4. Have undergone unilateral or bilateral implantation with a desired non-toric TECNIS IOL design (e.g., refractive or diffractive).
5. At least three months postoperative in the eligible eye.

EXCLUSION CRITERIA (ALL CRITERIA APPLY TO STUDY EYE)

1. Any medical or ocular history, in the opinion of the investigator, that may impact study procedures such as ocular trauma, pseudoexfoliation syndrome, retinal pigment degeneration, macular pathology, glaucoma, retinal disease, corneal disease, or corneal opacities.
2. Have any condition that may affect the eye's ability to fixate (e.g., amblyopia).
3. Have a history of corneal or intraocular surgery other than cataract surgery.
4. Using ocular or systemic medications known to interact with dilation drops.
5. Have a history of allergic reactions to dilation drops.
6. Have clinically significant pupil abnormalities (e.g., non-reactive, fixed, or abnormally shaped pupils).
7. Has an intraocular pressure of ≥ 21mm Hg before mydriasis.
8. Have a mydriatic pupil diameter of less than 6 mm.
9. Have participated in a clinical trial within 7 days prior to study enrollment.
10. An employee (e.g., Investigator, Coordinator, or Technician) or immediate family member (including partner, child, parent, grandparent, grandchild, or sibling) of an employee of the clinical site or study sponsor.
11. Currently pregnant or lactating.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As only one eye per subject will be enrolled in the study based on the eligibility criteria, up to approximately 80 subjects (40 by site) will be enrolled to obtain data on approximately 72 subjects (36 per site) to account for approximately 10% screen failure rate. All efforts will be made to enroll approximately 36 subjects per pre-study IOL group (i.e. 18 per site per pre-study IOL type).
  Approximately in total 36 subjects (18 per site) will be examined for each of the following two pre-study IOL groups.
  * Group 1: TECNIS refractive non-toric IOL models
  * Group 2: TECNIS diffractive non-toric IOL models
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Magnitude and Direction of IOL decentration and; Magnitude and Direction of IOL tilt. | One study visit
  The primary endpoints for this study will be:
  * Magnitude of IOL decentration relative to the visual axis through OCT (IOL Master 700) image analysis.
  * Direction of IOL decentration relative to the visual axis through OCT (IOL Master 700) image analysis.
  * Magnitude of IOL tilt relative to the visual axis through OCT (IOL Master 700) image analysis.
  * Direction of IOL tilt relative to the visual axis through OCT (IOL Master 700) image analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Surgical Vision Inc. Johnson and Johnson, Study Director — Sponsor GmbH
Locations (2):
- United States (2):
  - Empire Eye & Laser Center, Bakersfield, California
  - Jones Eye Center, Sioux City, Iowa

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu